CLINICAL TRIAL: NCT04537832
Title: ENVISION: Natural History Study of Infants and Children With Developmental and Epileptic Encephalopathies
Brief Title: Natural History Study of Infants and Children With Developmental and Epileptic Encephalopathies
Acronym: ENVISION
Status: Terminated | Type: Observational
Why Stopped: The ENVISION study has generated a robust data set that shows consistency in the seizure and non-seizure manifestations of SCN1A+ Dravet syndrome.
Sponsor: Encoded Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: ETX-DS-001
Record Dates: First submitted 2020-08-21; First posted 2020-09-03 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Dravet Syndrome
Keywords: severe myoclonic epilepsy; epilepsy; severe myoclonic epilepsy of infancy; SMEI; SCN1A related seizure disorder; epileptic encephalopathy; developmental and epileptic encephalopathies; DEE
MeSH Terms: conditions — Epilepsies, Myoclonic; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SCN1A-positive Dravet Syndrome: Participants aged between 6 and 60 months of age who have SCN1A-positive Dravet Syndrome. Clinical, neurocognitive, laboratory, the burden of disease, and health care resource utilization will be assessed.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
This is a multicenter, prospective, 2-year observational study in infants and children with developmental and epileptic encephalopathies (DEEs). The DEE currently being investigated is SCN1A-positive Dravet Syndrome.

DETAILED DESCRIPTION:
This prospective, longitudinal, natural history master protocol has been designed to define the seizure, neurodevelopmental, and behavioral characteristics of SCN1A-positive Dravet Syndrome in infants and children between 6 and 60 months. It will also explore the impact of the disease on the participant's parent/caregiver quality of life (QoL) and healthcare resource utilization (HCRU).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 6 months and 60 months.
* Confirmed SCN1A mutation.
* Normal development prior to onset of first seizure as defined by the Centers for Disease -Control and Prevention (CDC 2019).
* Onset of seizures between age 3 and 15 months, inclusive.

Exclusion Criteria:

* Copy number variant of SCN1A, including SCN1A microdeletion, if affecting other genes.
* SCN1A mutation present on both alleles.
* Known pathogenic or clinically suspected mutation in a seizure-associated gene besides SCN1A.
* Confirmed mutation in a gene besides SCN1A that is known to increase the severity of the seizure phenotype.
* Known gain-of-function genetic mutation, as defined by functional studies, including p.Thr226Met.
* History of notable developmental deficit that was evident prior to seizure onset.
* Known central nervous system structural abnormality as found on magnetic resonance imaging or computed tomography scan of brain.
* Currently taking or has taken for 6 or more consecutive weeks anti-seizure medications (ASMs) at a therapeutic dose that are contraindicated in SCN1A-positive Dravet Syndrome, including sodium channel blockers.
* Known concomitant genetic mutation or clinical comorbidity that potentially confounds typical Dravet phenotype.

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants and children aged between 6 and 60 months with SCN1A-positive Dravet Syndrome.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Seizure burden | Change from Baseline at 24 months
  Measured using monthly seizure frequency derived from seizure diaries.
Seizure freedom | Change from Baseline at 24 months
  Measured using the proportion of seizure-free days observed.
Use of anti-seizure medication(s) | Baseline through Month 24
  Measured using the incidence of anti-seizure medication usage observed during the 60 days leading up to each nominal visit.
Use of Special Diet | Change from Baseline at 24 months
  Measured using the incidence of ketogenic/high-fat diet usage observed during the 60 days leading up to each nominal visit.
Cognitive functioning | Change from Baseline at 24 months
  Measured using composite scores from 3 domains in the Bayley Scales of Infant and Toddler Development (3rd Edition) instrument. Domains include: (1) Cognitive; (2) Language; (3) Motor.
  Composite scores are normalized to a mean and SD of 100 and 15, respectively (range is not applicable as the scores are unbounded). Higher scores correspond to better outcomes compared to a normal population.
Behavioral and social functioning | Change from Baseline at 24 months
  Measured using raw scores from 2 domains in the Brief Infant Toddler Social Emotional Assessment. Domains include: (1) Problem; and (2) Competence.
  Domain raw scores range from 31 to 93 and 11 to 33 for the Problem and Competence domains, respectively. Higher Problem scores correspond to worse outcomes. Higher Competence scores correspond to better outcomes
Motor functioning | Baseline through Month 24
  Measured using categorical outcomes of 7 motor items adapted from the Bayley Scales of Infant and Toddler Development instrument and NorthStar Ambulatory Assessment. Motor milestones include: (1) Sit unassisted for 30 seconds; (2) Walk with assistance; (3) Stand alone; (4) Walk alone; (5) Walk upstairs; (6) Run with Coordination; and (7)Jump forward.
Incidence of Adverse Events | Baseline through Month 24
  Measured using the incidence of adverse events and serious adverse events (broken down by preferred term) observed during the study.
Overall survival | Baseline through Month 24
  Measured using the incidence of death observed by a given time point during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Rico, M.D., Ph.D, Study Director — Encoded Therapeutics
Locations (16):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nicklaus Children's Hospital, Miami, Florida
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Abigail Wexner Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Multicare Institute for Research and Innovation, Tacoma, Washington
- Austin Hospital - Melbourne Brain Centre, Heidelberg, Victoria, Australia
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari i Politècnic La Fe, Valencia
- Queen Elizabeth Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Plan is undecided